CLINICAL TRIAL: NCT02998073
Title: A Multiple Biomarker Approach to Investigating Psychosocial Intervention Treatment Response in Justice-Involved Youth With Conduct Disorder
Brief Title: Investigating Psychosocial Intervention Treatment Response in Justice-Involved Youth With Conduct Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Ontario Mental Health Foundation (Other Government)
Responsible Party: Principal Investigator, Nathan Kolla, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0702016
Record Dates: First submitted 2016-12-14; First posted 2016-12-20 (Estimated); Last update posted 2021-08-16 (Actual); Status verified 2021-08

CONDITIONS: Conduct Disorder
MeSH Terms: conditions — Conduct Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conduct Disorder (Experimental): Participants are justice-involved youth with conduct disorder. Participants will receive Stop, Now and Plan (SNAP) psychosocial intervention.
  Interventions: Behavioral: Stop, Now and Plan
- Control (No Intervention): Participants are healthy males. Participants receive no intervention.

INTERVENTIONS:
Behavioral: Stop, Now and Plan — SNAP program was developed to target justice-involved youth (6 years and older) who have problems with aggression, CD, and/or gang affiliation. SNAP focuses on engaging youth in interesting and creative learning modules by providing real life scenarios designed to improve self-control, impulsive behaviors, decision-making skills, and pro-social skills. SNAP treatment is delivered over a 13-week period.
  Arms: Conduct Disorder

SUMMARY:
This research focuses on youth with conduct disorder (CD), and a history of violence. CD is a youth neurodevelopmental disorder that is commonly associated with criminality. Although psychosocial interventions that address impulsivity and self-control have been shown to be effective at helping promote prosocial behavior in patients with CD, the biological changes that occur as a result of treatment are not well understood. This study will explore changes in the brain function of the anterior cingulate cortex (ACC) in response to a common psychosocial intervention (Stop, Now and Plan). This study will contribute to our understanding of biological mechanisms involved in therapeutic gains among children with behavioural problems and youth offenders; therefore, it will inform further development of treatment programs for children/youth with impulsive behaviours.

DETAILED DESCRIPTION:
CD is a youth-limited neurodevelopmental disorder characterized by impulsivity and dysfunctional social behavior. CD is associated with increased risks of mortality, lower educational and occupational achievement, criminal behavior and other psychosocial difficulties, and hence presents a significant burden to society. Impulsivity is a prominent predictor of violence in CD. Treatment programs targeting impulsivity in CD have been shown to be effective at increasing pro-social functioning in CD, but the biological mechanisms that underpin these therapeutic gains are not well understood. Past research suggests that the ACC play a role in CD and impulsivity. This study explores biological and behavioral changes in response to Stop, Now and Plan (SNAP), a validated 13-week psychosocial intervention addressing impulsivity and self-control in youth.

The main hypotheses are:

(1) CD youth who respond to SNAP treatment will exhibit greater post-treatment ACC activation during an fMRI imaging task compared with their baseline, pre-treatment ACC activation.

The secondary hypotheses are:

(1) CD youth will exhibit lower ACC activation at baseline during an fMRI imaging task compared with the baseline ACC activation exhibited by typically developing youth.

ELIGIBILITY:
Inclusion Criteria (SNAP Treatment Group):

- Historical diagnosis of CD as per the K-SADS, which will be corroborated by DSM-5 criteria obtained by clinical assessment, and a CBCL, externalizing sub-score of 70 and above.

Inclusion Criteria (SNAP Control Group)

* No history of psychiatric illness as assessed by the Kiddi - Schedule for Affective Disorders and Schizophrenia Present and Lifetime version (K-SADS)
* No history of criminal justice system involvement.

Exclusion Criteria (ALL Groups):

* Serious, unstable medical condition that precludes safe participation in the study
* History of neurological or endocrine disorder
* Any contraindication to safe MRI scanning, including claustrophobia
* Psychotic or bipolar disorder
* Current drug use measured by urinalysis
* Full-scale IQ of 80 or lower (cut-off for borderline intellectual functioning) measured using the Wechsler Abbreviated Scales of Intelligence - 2nd Edition (WASI-II)

Ages: 6 Years to 11 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2020-02-05 (Actual); Study Completion 2021-08-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline: blood-oxygen-level dependent (BOLD) activation of anterior cingulate cortex as measured by functional magnetic resonance imaging | Measured before and after the 13-week program
  Difference in ACC BOLD activation to commission errors (contrast of BOLD response during commission errors vs. BOLD response during correct hits) will be tested using a 2 (Session: pre-SNAP vs. post-SNAP) × 2 (Group: treatment responders vs. non-treatment responders) within subject, mixed model analysis of covariance (ANCOVA), controlling for the effect of age, to investigate the two-way interaction between session and group. (Note: Commission errors compose a measure produced by the Go/No-Go task.)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Kolla, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research